CLINICAL TRIAL: NCT00015470
Title: Diagnostic Evaluation of Patients With Neuromuscular Diseases
Brief Title: Diagnostic Evaluation of Patients With Neuromuscular Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010149; 01-N-0149
Record Dates: First submitted 2001-04-19; First posted 2001-04-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-05-10

CONDITIONS: Neuromuscular Disease
Keywords: Myopathy; Dystrophy; Neuropathy; Muscle Weakness; Muscle Cramps and Pains; Neuromuscular Disorders
MeSH Terms: conditions — Neuromuscular Diseases; Muscular Diseases; Muscle Weakness; Muscle Cramp; Pain

SUMMARY:
The objectives of this protocol are to: 1) screen patients with various neuromuscular disorders and facilitate their entry into appropriate research protocols; 2) help resolve puzzling diagnostic neuromuscular problems and train fellows in the evaluation and treatment of Neuromuscular Diseases; and 3) provide follow up to patients who finished their participation in a previous study but they are not currently entered in another research protocol. No investigational treatments will be performed on this protocol but the tissues collected can be used for future research studies.

DETAILED DESCRIPTION:
The objectives of this protocol are to: 1) screen patients with various neuromuscular disorders and facilitate their entry into appropriate research protocols; 2) help resolve puzzling diagnostic neuromuscular problems and train fellows in the evaluation and treatment of Neuromuscular Diseases; and 3) provide follow up to patients who finished their participation in a previous study but they are not currently entered in another research protocol. No investigational treatments will be performed on this protocol but the tissues collected can be used for future research studies.

ELIGIBILITY:
* INCLUSION CRITERIA:

Research patients will be studied under this protocol if they fulfill the following criteria:

Have an identifiable neuromuscular disorder that may be suitable for a specific current or future protocol;

Present a diagnostic puzzle in spite of the previously performed diagnostic work-up;

Have unusual manifestation of a more usual neuromuscular disease;

Have a disorder useful for teaching purposes.

Patients should be referred by a physician who will continue their care after our evaluation. A report of the patients' visit and tests, along with suggestions or recommendations will be sent to each referring physician. There is a wide spectrum of neuromuscular diseases to be studied, among them are: peripheral neuropathies, myopathies, dystrophies, myasthenia, stiff person syndrome, muscle cramps, myotonias, motor neuron diseases, post-polio syndrome, and certain demyelinating disorders affecting both the central and the peripheral nervous system.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500
Dates: Start 2001-04-16; Study Completion 2007-05-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States